## Inflammation in Women with Urgency Urinary Incontinence Treated with Anticholinergics

**Version Date: 7/28/2022** 

ID: 2018P000980

Study Name: Inflammation in Women with Urgency Urinary Incontinence Treated with

Anticholinergics

PI Name: Dr. Vatche A. Minassian

Prepared by: Alexa Courtepatte, B.S., Research Assistant

**Specific Aim 1:** To assess inflammatory markers in urine and serum before and after a 6-week treatment course with anticholinergies.

**Specific Aim 2:** To determine the role of the urinary microbiome in relation to inflammation before and after a 6-week treatment course with anticholinergics.

**Study Population:** This study is a prospective pilot of women who have a diagnosis of urge urinary incontinence (UUI) and present to the BWH Urogynecology Clinics in Boston or Foxborough. This study enrolled 20 women offered standard of care anticholinergic treatment for 6 weeks.

**Statistical Methods:** Demographic and clinical characteristics were summarized with the absolute count and percent of categorical variables and median and interquartile range of continuous variables. No comparison was made as demographic and clinical characteristics did not change in follow-up period.

Plasma and combined (baseline and follow-up) urine cytokines were summarized using median and interquartile range.

Urine cytokines at baßseline and follow-up were tested for normality using Shapiro-Wilks test for normality. The data were found to be non-normal and thus were summarized using median and interquartile range. Urine cytokines were compared from baseline to follow-up for most patients (only 13 of the 20 patients returned for follow-up) using t-test of Wilcoxon rank sum. P value of <0.05 was considered significant.